CLINICAL TRIAL: NCT02282046
Title: Diabetes Effects on Long-Term Implant Survival and Success
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-444H; R01DE023518 (NIH)
Record Dates: First submitted 2014-09-15; First posted 2014-11-04 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; dental implant
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non-diabetic group: patients without diagnosed type 2 diabetes, having an HbA1c level below 6.0%
- type 2 diabetes group: patients diagnosed with type 2 diabetes of over 1 year duration.

SUMMARY:
This study is designed to understand the impact of glycemic control in patients with type 2 diabetes on dental implants under long-term function. It is hypothesized that poor glycemic control will not have significant effects on implant-related outcomes over longer periods of time.

DETAILED DESCRIPTION:
This single-center prospective observational cohort study seeks to clarify the role of glycemic control as a risk determinant for survival of dental implants and biologic complications of dental implant therapy in patients with type 2 diabetes. Long-term implant stability and implant-related complications will be assessed in relation to glycated hemoglobin levels over time in poorly-controlled and well-controlled diabetics and in non-diabetic participants.

Primary: To determine the impact of glycemic control in type 2 diabetes patients on implant-related biologic complications, integration and survival for dental implants under long-term functional loading (>1 year).

Secondary: To examine these associations relative to long-term effects of sub-optimal glycemic control on two different anatomic/restorative schemes (fixed partial or removable complete) Outcomes: Assessments include implant survival, implant-related biologic complications and resonance frequency analysis as a measure of implant stabilization. Outcomes will be analyzed relative to glycated hemoglobin levels (HbA1c) taken at 6-month intervals over the course of the study.

The total study population will consist of 163 participants who will be followed for at least 2 years. This will include enrolling from a group of 141 patients who have previously received implant therapy as part of short-term assessments regarding diabetes.

In addition, the study plans to enroll 42 participants who would benefit from implant supported denture therapy as done in the prior studies. These participants will be classified into 3 separate groups depending on the A1C reading at time of implant placement. The criteria being followed for the groups are HbA1c< 6.0% (non-diabetic), 6.0%<HbA1c<8.0% (well controlled diabetic) and 8.0%<HbA1c<12.0% (poorly controlled diabetic).

A review of the potential participant's health is completed at the time of screening. The implant surgeon will determine if a patient is healthy for surgery with no anticipated health complications. If a health concern is evident that precludes implant placement, the patient will be excluded from study participation.

The age requirement for the study is 25 years of age or older. It is expected that most participants will be 50 years and over due to the specific clinical requirements for the treatment being followed. Individuals of any gender, race, and ethnicity may participate in this study. Most patients live locally in San Antonio, TX and some are from the surrounding cities.

ELIGIBILITY:
Inclusion Criteria:

* • Provide signed and dated informed consent form.

  * Willing to comply with all study procedures and be available for the duration of the study.
  * For participants with existing implant therapy: participated in either of two previous observational diabetes-implant studies that monitored implant outcomes and glycemic levels as conducted by Dr. Oates [IRB study #s: HSC20070499H & HSC20080156H].
  * For edentulous participants without existing implant therapy: Diagnosis of type 2 diabetes mellitus occurring more than 1 year prior to enrollment (self-reported and verified with physician report, test results, and/or treatment record) or healthy, non-diabetic with a HbA1c < 6.0%, or either FPG < 100 mg/dl or an OGTT < 140 mg/dl (2 hr) within 11 months prior to surgery; participants must have complete maxillary and mandibular dentures determined to be clinically acceptable by study dentists; and must have an identified need for 2-implant supported mandibular overdenture using standard diameter Straumann 4.1 mm implants.
  * Male or female, aged 25 to 99.
  * HbA1c <12%.
  * Women of reproductive potential must report a negative urine pregnancy test within 2 weeks of enrollment in study, and agree to use highly effective contraception during study period. Acceptable methods of birth control include abstinence, oral contraceptives, the contraceptive patch, the contraceptive ring, and condoms.

Exclusion Criteria:

* Medical condition, laboratory finding, or physical exam finding that precludes implant placement or therapy (including cardiovascular, hepatic, renal, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, autoimmune, or psychiatric disorders).

  * Current medications or history of treatment known to have an effect on bone turnover, including: calcitonin, systemic steroids, bisphosphonates, estrogen or progesterone therapy.
  * Presence of acute untreated oral infections or inflammatory lesions.
  * History of HIV infection, Hepatitis B or C as determined by patient report or medical record.
  * Self-reported history of illicit drug use or alcohol abuse (Appendix D).
  * Implant site has had bone grafting procedures using autogenic or allogenic materials less than one year prior to placement, or requires bone grafting in conjunction with implant placement.
  * Implant site has had alloplastic grafting procedures.
  * Presence of a disease that affects bone metabolism, such as but not limited to: hyperthyroidism, hyperparathyroidism, congenital connective tissue disorders (e.g., osteogenesis imperfecta), or Paget's disease.
  * Participation in a clinical study that may interfere with participation in this study during the implant surgical phase and healing 4 months following placement.
  * Self-reported current tobacco use
  * Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will include those edentulous patients benefiting from mandibular implant overdenture support. It may include those already being followed in a similar study or patients newly receiving dental implants. It will also include type 2 diabetes patients who received dental implant therapy as part of a previous study on the impact of glycemic control.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2014-05; Primary Completion 2018-05-15 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
implant complications | at an anticipated average of 5 years following placement
  long-term clinical evaluations will be performed every 6 months.
  biologic complications assessed will include signs of infection, inflammation, bone loss, and implant failure.

SECONDARY OUTCOMES:
resonance frequency analysis | at an anticipated average of 5 years following placement
  implant stability will be measured at 6 month intervals using resonance frequency analysis.

CONTACTS AND LOCATIONS:
Overall Officials: thomas oates, dmd, phd, Principal Investigator — University of Texas Health Science Ctr a
Locations (1):
- University of Texas Health Science Center At San Antonio, San Antonio, Texas, United States